CLINICAL TRIAL: NCT05196958
Title: Interest of GLP1 Analogues (aGLP1) in Overweight Type 2 Diabetic Patients With Chronic Inflammatory Bowel Disease (IBD)
Brief Title: Interest of GLP1 Analogues in Overweight Type 2 Diabetic Patients With Chronic Inflammatory Bowel Disease
Acronym: DiagMICI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DiagMICI
Record Dates: First submitted 2021-12-30; First posted 2022-01-19 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Inflammatory Bowel Diseases; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Inflammatory Bowel Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GLP1 analogues (Experimental): This cohort study has 2 phases: an observation phase to collect all initial clinical and biological parameters and an intervention phase (prescription of GLP1 analogues) of 6 months including a visit at 3 and 6 months.
  Interventions: Other: GLP1 analogues

INTERVENTIONS:
Other: GLP1 analogues — This cohort study has 2 phases: an observation phase to collect all initial clinical and biological parameters and an intervention phase (prescription of GLP1 analogues) of 6 months including a visit at 3 and 6 months.

SUMMARY:
The risk of type 2 diabetes appears to be higher in patients with chronic inflammatory diseases, including chronic inflammatory bowel disease (IBD). IBD is a group of inflammatory diseases that includes mainly Crohn's disease and ulcerative colitis.

Although the majority of IBD patients are not overweight, the prevalence of obesity in this population remains significant, estimated at 15 to 40%. It has been shown that obesity can impact the response to therapies used in IBD as well as the clinical course of the disease:

1) plasma concentrations of immunomodulatory therapies are often lower in the obese compared to those with a normal Body Mass Index (BMI) with a lower dose per kg of the administered drug as well as an acceleration of drug clearance.

2nd) Surgical management of IBD is associated with a higher risk of peri- and post-operative complications in obese patients, including an increase in operating time, bleeding risk, length of hospital stay and percentage of post-operative infections.

3e) Finally, obesity seems to have a negative impact on the clinical course of IBD, with a correlation between an increase in BMI and an increase in the number of hospitalizations, the number of follow-up consultations and the need for therapeutic escalation.

One of the common pathophysiological explanations between IBD and metabolic syndrome (including type 2 diabetes and obesity), would involve metabolites in the gut that are modulated by the gut microbiota.

Glucagon-Like Peptide 1 (aGLP1) analogues are a new class of injectable antidiabetic drugs that have revolutionized the management of type 2 diabetes. They include exenatide, lixisenatide, liraglutide, dulaglutide and semaglutide. They combine an effect on glycemic control but also usually a weight loss. In some countries, they are used in non-diabetic obese patients, with a weight loss of up to -10 to -15%. These molecules bind to GLP1 receptors, stimulate insulin secretion when blood glucose levels are high, decrease glucagon secretion, slow gastric emptying and stimulate satiety. In addition to glycemic control, weight reduction is most often associated.

In addition, some aGLP1s have been shown to reduce cardiovascular events in diabetics. They are well tolerated, but their side effects are mainly digestive, such as nausea, vomiting and sometimes diarrhea. These problems occur in about 20% of cases, most often after the first injection, with vomiting requiring permanent cessation of treatment. Most often they gradually subside, spontaneously or after symptomatic treatment, and allow titration of the drug.

Due to the lack of studies and possible intestinal effects, aGLP1 is not recommended in cases of severe gastrointestinal disease, and therefore in cases of IBD, although it is not contraindicated.

The main objective of this study is to test the interest of these GLP1 analogues in type 2 diabetics with IBD, who are overweight and whose glycemic target is not reached. The expected benefit is to facilitate diabetes control and weight loss in this population. The second objective is to monitor the occurrence of adverse events in this population with the different GLP1 analogues used.

ELIGIBILITY:
* Patients between 18 and 75 years of age
* Patients with inflammatory bowel disease (Crohn's disease (CD) or ulcerative colitis (UC))
* Patient with poorly controlled type 2 diabetes (defined as deviation from the set glycemic target of more than 1% HbA1c)
* Patient with a BMI ≥ 25 kg/m2
* For women of childbearing age: effective contraception* during treatment and up to 5 weeks after discontinuation

  * Any contraceptive method used regularly and appropriately that has a low failure rate (i.e., less than 1% per year)
* Patient enrolled in a health insurance plan
* Francophone patient
* Patient with free, informed, written consent

Exclusion Criteria:

* Patient with a personal or family history of medullary thyroid cancer
* Patient with an active cancer
* Patient with a history of acute or chronic pancreatitis
* Patients with a history of hypersensitivity to GLP1 analogues (or to any other component of the product)
* Patient with a history of severe GI intolerance to GLP-1 receptor agonists
* Patient already included in a risky interventional research protocol (RIPH1)
* Pregnant or breastfeeding women
* Patients with congestive heart failure New York Heart Association (NYHA) class IV
* Patient with end-stage renal disease
* Patients with clinically significant sustained elevation of resting heart rate
* Patient with anti-GAD antibodies in a previous workup at inclusion
* Patient under guardianship or curatorship
* Patient under court protection
* Patient deprived of liberty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2024-01-14 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycemic control | Month 6
  This outcome corresponds to the Change in HbA1c at 3 and 6 months compared with baseline at initiation of therapy.
Weight loss | Month 6
  This outcome corresponds to the weight reducation at 3 and 6 months compared to baseline.

SECONDARY OUTCOMES:
Tolerance of GLP1 analogues after 3 months of treatment | Month 3
  This outcome corresponds to th number of serious and non-serious adverse events after 3 months of treatment with aGLP1.
Tolerance of GLP1 analogues after 6 months of treatment tolerance of GLP1 analogues after 3 and 6 months of treatment | Month 6
  This outcome corresponds to the number of serious and non-serious adverse events after 6 months of treatment with aGLP1.
Quality of life after 3 months of treatment | Month 3
  This outcome corresponds to the Quality of life of patients according to the Inflammatory Bowel Disease Questionnaire score. It includes 32 items in four domains: digestive symptoms (10 items), systemic symptoms (5 items), emotional disorders (12 items), social function (5 items). Each item is measured using the Likert technique. For each item, the interviewer presents a set of 7 statements describing an attitude. To each degree of agreement, a numerical value (from 1 to 7) is attached. In this way, by adding the individual scores, a total numerical value can be calculated. The total score ranges from 32 to 224, the higher the score the better the quality of life. This index has been validated and is correlated with the different disease activity scores.
Quality of life after 6 months of treatment | Month 6
  This outcome corresponds to the Quality of life of patients according to the Inflammatory Bowel Disease Questionnaire score. It includes 32 items in four domains: digestive symptoms (10 items), systemic symptoms (5 items), emotional disorders (12 items), social function (5 items). Each item is measured using the Likert technique. For each item, the interviewer presents a set of 7 statements describing an attitude. To each degree of agreement, a numerical value (from 1 to 7) is attached. In this way, by adding the individual scores, a total numerical value can be calculated. The total score ranges from 32 to 224, the higher the score the better the quality of life. This index has been validated and is correlated with the different disease activity scores.
Impact of aGLP1 on the treatment already in place to regulate blood glucose | Month 6
  This outcome corresponds to the reduction in number/dose of anti-diabetic medications or daily insulin dose.

CONTACTS AND LOCATIONS:
Overall Officials: Adela VOICAN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Dregan A, Charlton J, Chowienczyk P, Gulliford MC. Chronic inflammatory disorders and risk of type 2 diabetes mellitus, coronary heart disease, and stroke: a population-based cohort study. Circulation. 2014 Sep 2;130(10):837-44. doi: 10.1161/CIRCULATIONAHA.114.009990. Epub 2014 Jun 26. PMID 24970784
- [Background] Jess T, Jensen BW, Andersson M, Villumsen M, Allin KH. Inflammatory Bowel Diseases Increase Risk of Type 2 Diabetes in a Nationwide Cohort Study. Clin Gastroenterol Hepatol. 2020 Apr;18(4):881-888.e1. doi: 10.1016/j.cgh.2019.07.052. Epub 2019 Aug 5. PMID 31394285
- [Background] Singh S, Dulai PS, Zarrinpar A, Ramamoorthy S, Sandborn WJ. Obesity in IBD: epidemiology, pathogenesis, disease course and treatment outcomes. Nat Rev Gastroenterol Hepatol. 2017 Feb;14(2):110-121. doi: 10.1038/nrgastro.2016.181. Epub 2016 Nov 30. PMID 27899815
- [Background] Seminerio JL, Koutroubakis IE, Ramos-Rivers C, Hashash JG, Dudekula A, Regueiro M, Baidoo L, Barrie A, Swoger J, Schwartz M, Weyant K, Dunn MA, Binion DG. Impact of Obesity on the Management and Clinical Course of Patients with Inflammatory Bowel Disease. Inflamm Bowel Dis. 2015 Dec;21(12):2857-63. doi: 10.1097/MIB.0000000000000560. PMID 26241001
- [Background] Hicks G, Abdulaal A, Slesser AAP, Mohsen Y. Outcomes of inflammatory bowel disease surgery in obese versus non-obese patients: a meta-analysis. Tech Coloproctol. 2019 Oct;23(10):947-955. doi: 10.1007/s10151-019-02080-0. Epub 2019 Sep 17. PMID 31531732
- [Background] Pavelock N, Masood U, Minchenberg S, Heisig D. Effects of obesity on the course of inflammatory bowel disease. Proc (Bayl Univ Med Cent). 2019 Feb 1;32(1):14-17. doi: 10.1080/08998280.2018.1542887. eCollection 2019 Jan. PMID 30956572
- [Background] Verdugo-Meza A, Ye J, Dadlani H, Ghosh S, Gibson DL. Connecting the Dots Between Inflammatory Bowel Disease and Metabolic Syndrome: A Focus on Gut-Derived Metabolites. Nutrients. 2020 May 15;12(5):1434. doi: 10.3390/nu12051434. PMID 32429195
- [Background] Nauck M, Frid A, Hermansen K, Shah NS, Tankova T, Mitha IH, Zdravkovic M, During M, Matthews DR; LEAD-2 Study Group. Efficacy and safety comparison of liraglutide, glimepiride, and placebo, all in combination with metformin, in type 2 diabetes: the LEAD (liraglutide effect and action in diabetes)-2 study. Diabetes Care. 2009 Jan;32(1):84-90. doi: 10.2337/dc08-1355. Epub 2008 Oct 17. PMID 18931095
- [Background] O'Neil PM, Birkenfeld AL, McGowan B, Mosenzon O, Pedersen SD, Wharton S, Carson CG, Jepsen CH, Kabisch M, Wilding JPH. Efficacy and safety of semaglutide compared with liraglutide and placebo for weight loss in patients with obesity: a randomised, double-blind, placebo and active controlled, dose-ranging, phase 2 trial. Lancet. 2018 Aug 25;392(10148):637-649. doi: 10.1016/S0140-6736(18)31773-2. Epub 2018 Aug 16. PMID 30122305
- [Background] Astrup A, Rossner S, Van Gaal L, Rissanen A, Niskanen L, Al Hakim M, Madsen J, Rasmussen MF, Lean ME; NN8022-1807 Study Group. Effects of liraglutide in the treatment of obesity: a randomised, double-blind, placebo-controlled study. Lancet. 2009 Nov 7;374(9701):1606-16. doi: 10.1016/S0140-6736(09)61375-1. Epub 2009 Oct 23. PMID 19853906
- [Background] Zatorski H, Salaga M, Fichna J. Role of glucagon-like peptides in inflammatory bowel diseases-current knowledge and future perspectives. Naunyn Schmiedebergs Arch Pharmacol. 2019 Nov;392(11):1321-1330. doi: 10.1007/s00210-019-01698-z. Epub 2019 Jul 29. PMID 31359088